CLINICAL TRIAL: NCT01912820
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled Two-Arm Study of Quercetin and Green Tea to Enhance the Bioavailability of Green Tea Polyphenols in Men Scheduled for Prostatectomy
Brief Title: Effect of Quercetin on Green Tea Polyphenol Uptake in Prostate Tissue From Patients With Prostate Cancer Undergoing Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12-000886; NCI-2013-01153 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R03CA171583 (NIH)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tea; Quercetin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (quercetin, green tea extract) (Experimental): Patients receive GT extract PO BID and quercetin PO BID for 3-6 weeks before undergoing prostatectomy.
  Interventions: Dietary Supplement: green tea extract; Drug: quercetin; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis
- Arm II (GT extract, placebo) (Placebo Comparator): Patients receive GT extract PO BID and placebo PO BID for 3-6 weeks before undergoing prostatectomy.
  Interventions: Dietary Supplement: green tea extract; Other: placebo; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Dietary Supplement: green tea extract — Given PO
  Other Names: green tea polyphenols
Drug: quercetin — Given PO
  Other Names: C.I. natural yellow 10
  Arms: Arm I (quercetin, green tea extract)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (GT extract, placebo)
Procedure: therapeutic conventional surgery — Undergo prostatectomy
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized pilot phase I trial will evaluate if quercetin enhances the uptake of green tea polyphenols in the prostate tissue of men taking green tea extract and undergoing radical prostatectomy. Side effects of green tea extract and quercetin in combination with green tea extract will also be evaluated. In preclinical studies, green tea polyphenols have anticancer and cancer preventative effects in a number of malignancies. Likewise, in preclinical studies quercetin was found to enhance the anticancer effects of green tea. This trial is designed to translate these findings forward in a short-term human intervention trial.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the prostate tissue concentration of epigallocatechin gallate (EGCG), epicatechin gallate (ECG) and quercetin and their methylated metabolites in men scheduled for prostatectomy and consuming green tea (GT)extract (N=15) or GTextract with quercetin (N=15) for 3 weeks prior to prostatectomy.

II. To determine the concentration of EGCG, ECG, epigallocatechin (EGC), epicatechin (EC) and quercetin and the methylated metabolites in plasma collected before (T=0) and two hours (T=2) after the intake of the morning dose of GTextract and placebo or GTextract with quercetin during the third week of intervention.

III. To determine the effect of GTextract/quercetin intervention on reducing the enzyme activity and protein and gene expression of catechol-O-methyltransferase (COMT) and deoxyribonucleic (DNA) (cytosine-5) methyltransferase 1 (DNMT1) as well as protein and gene expression of multidrug resistance transport protein 1 (MRP1) in prostate tissue collected in specific aim 1 and COMT activity in erythrocytes from blood collected at baseline and week 3.

IV. To determine the inter-individual variation in genotype of COMT in buffy coat DNA.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive GT extract orally (PO) twice daily (BID) and quercetin PO BID for 3-6 weeks before undergoing prostatectomy.

ARM II: Patients receive GT extract PO BID and placebo PO BID for 3-6 weeks before undergoing prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects consent to participate in the trial
* The subject has a diagnosis of adenocarcinoma of the prostate
* The subject is scheduled to undergo radical prostatectomy
* The subject agrees to stop consuming tea or tea-containing products and quercetin supplements throughout the entire intervention period except for the green tea extract and quercetin provided during study intervention

Exclusion Criteria:

* History of hepatitis or liver dysfunction
* Ongoing alcohol abuse
* Significant medical or psychiatric conditions that would make the patient a poor protocol candidate
* Prior sensitivity or allergic reaction to tea, tea products or tea and quercetin supplements
* Allergies to multiple food items or nutritional supplements
* Taking luteinizing hormone-releasing hormone (LHRH) agonists, androgen receptor blocking agents, finasteride, or has undergone bilateral orchiectomy

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Green tea polyphenols, quercetin and their metabolite concentration in blood and prostate tissue | On the day of surgery
  Means and standard deviation will be calculated and the statistical difference between treatment with GTextract + quercetin compared to GTextract + placebo will be determined using Student's t-test computed by one-way analysis of variance models.

SECONDARY OUTCOMES:
Protein and gene expression of COMT in prostate tissue | Day of surgery
Protein and gene expression of DNMT1 in prostate tissue | Day of surgery
Protein and gene expression of MRP1 in prostate tissue | Day of surgery
COMT activity in red blood cells | Week 3
Genotype of COMT (high [H]/H, low [L]/L or H/L) | Week 3
  Gene-association analyses will be conducted for COMT polymorphic variants within each intervention group using SAS Genetics, version 9.1

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Henning, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Veterans Administration Los Angeles Healthcare System, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, Los Angeles, California